CLINICAL TRIAL: NCT02545387
Title: Hepatitis C Virus in Neutrophil Granulocyte Progenitor Cells
Status: Withdrawn | Type: Observational
Why Stopped: Logistical problems
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: HCV-KM
Record Dates: First submitted 2015-07-29; First posted 2015-09-10 (Estimated); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — serum liver tissue bone marrow
Oversight: Data Monitoring Committee: No

SUMMARY:
Patients with hepatitis C show impaired neutrophil function. It is not known whether this is a direct of an indirect phenomenon. Using bone marrow biopsies from patients with hepatitis C it is possible to see whether neutrophil granulocyte progenitors are already infected with hepatitis C.

DETAILED DESCRIPTION:
Neutrophil granulocytes are important components of the innate immune system and pioneers in the fight against both fungal and bacterial infections. If pathogens enter the body, they are marked as foreign by antibodies and the complement system. Afterwards receptors on the neutrophils recognize and bind on these foreign substances to make them harmless. This process is called phagocytosis. Hepatitis C virus (HCV) and neutrophils are rarely associated. The HCV belongs to the Flaviviridae. It is a single-stranded, enveloped RNA virus with a positive polarity, which cause chronic hepatitis C (CHC) in approximately 170 million people worldwide. Subsequently, such an infection leads to liver cirrhosis and carcinoma in a significant proportion of patients. The virus infects mainly hepatocytes, but extrahepatic replication has also been shown. HCV usually enters the cell through receptor-mediated endocytosis (claudin-1, cluster of differentiation (CD)81, occludin and scavenger receptor 1), before it abuses the cell's own infrastructure for the viral protein synthesis.

The aim of this study is to determine neutrophil function in chronic hepatitis C infected patients. Furthermore the investigators want to examine if neutrophils or their precursor cells are infected with HCV and if this leads to their dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* chronic hepatitis C
* Genotype 1-4

Exclusion Criteria:

* acute hepatitis C

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: cells and tissue from patients with chronic hepatitis C virus infection
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
viral RNA | day 1
  hepatitis C virus RNA

SECONDARY OUTCOMES:
neutrophil phagocytic capacity | day 1
  function of neutrophil granulocytes in hepatitis C patients
hepatitis C virus proteins | day 1
  presence of hepatitis C virus proteins in neutrophils

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Stadlbauer, Principal Investigator — Medical University of Graz
Locations (1):
- Department of Internal Medicine, Medical University of Graz, Graz, Austria